CLINICAL TRIAL: NCT01296620
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Intravenous (IV) Ulimorelin Administered Post-Operatively to Accelerate Recovery of Gastrointestinal (GI) Motility in Subjects Who Have Undergone Partial Bowel Resection
Brief Title: Ulimorelin Study of Efficacy and Safety (ULISES 008)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tranzyme, Inc. (Industry)
Collaborators: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TZP-101-CL-P008; 2010-023229-38 (EudraCT Number)
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Gastrointestinal Dysmotility
MeSH Terms: interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Experimental 1 (Experimental)
  Interventions: Drug: Ulimorelin Intravenously (IV)
- Experimental 2 (Experimental)
  Interventions: Drug: Ulimorelin Invtravenously (IV)
- Placebo (Placebo Comparator)
  Interventions: Drug: 5% dextrose in water

INTERVENTIONS:
Drug: Ulimorelin Intravenously (IV) — 160 µg/kg daily (QD)
  Arms: Experimental 1
Drug: Ulimorelin Invtravenously (IV) — 480 µg/kg daily (QD)
  Arms: Experimental 2
Drug: 5% dextrose in water — Placebo
  Arms: Placebo

SUMMARY:
Post-operative administration of ulimorelin is expected to reduce time to recovery of Gastrointestinal (GI) function in patients who have undergone partial large bowel resection

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 to 80 years of age, inclusive
* Scheduled to undergo open bowel resection with colonic anastomosis
* For women who can potentially become pregnant a pregnancy test at screening and admission must be negative

Exclusion Criteria:

* Weight more than 200kg (441 pounds)
* Pregnant or breastfeeding
* Known history of drug or alcohol abuse within the previous year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Recovery of GI Function | up to 7 days of dosing or until hospital discharge

SECONDARY OUTCOMES:
Ancillary GI Functions | up to 7 days of dosing or hospital discharge

CONTACTS AND LOCATIONS:
Locations (50):
- United States (26):
  - Glendale Memorial Hospital, Glendale, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Univ. of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Palo Alto VA Health Care Ctr, Palo Alto, California
  - Citrus Memorial Hospital, Inverness, Florida
  - Pensacola Research Consultants, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - ARS Clinical Trials, Powder Springs, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - NOLA CVT Surgery, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CRC of Jackson, Jackson, Mississippi
  - Mount Sinai Hospital, New York, New York
  - Sanford Medical Center, Fargo, North Dakota
  - Kaiser Permanente Northwest, Clackamas, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Forbes Regional Hospita, Monroeville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Southwest Surgical Associates, Houston, Texas
  - VCU Medical Center, Richmond, Virginia
  - MultiCare Research Institute, Tacoma, Washington
- Bulgaria (5):
  - UMHAT Emergency Medicine, Sifua
  - MHAT Tokuda Hospital Sofia, Sofia
  - Military Medical Academy, Sofia
  - UMHAT Tzaritza Yoanna ISUL, Sofia
  - UMHAT St. Marina, Varna
- Czechia (7):
  - FN Brno, Brno
  - St. Anne's University Hospital, Brno
  - Hospital Jihlava, Jihlava
  - Hospital Liberec, Liberec
  - FN Olomouc, Olomouc
  - Fakutni Thomayerova nemocnica, Prague
  - University Hospital Bulovka, Prague
- France (4):
  - CHU Avicenne, Bobigny
  - Hopital Beaujon, Clichy Paris
  - CHRU Lille, Lille
  - CHU Rouen, Hopital Charles Nicolle, Rouen
- Lithuania (6):
  - Kaunas Clinical Hospital No. 2, Kaunas
  - Kaunas Medical University Clinics, Kaunas
  - Republican Klaipeda Hospital, Klaipėda
  - Klaipeda Hospital, Klaipėda
  - Institute of Oncology at Vilnius University, Clinic of Surgery, Vilnius
  - Vilnius City Univ. Hospital Clinic of Surgery, Vilnius
- Romania (2):
  - Institute regional de Gastroenterologie si Hepatologie, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta, Oradea

REFERENCES:
- [Derived] Shaw M, Pediconi C, McVey D, Mondou E, Quinn J, Chamblin B, Rousseau F. Safety and efficacy of ulimorelin administered postoperatively to accelerate recovery of gastrointestinal motility following partial bowel resection: results of two randomized, placebo-controlled phase 3 trials. Dis Colon Rectum. 2013 Jul;56(7):888-97. doi: 10.1097/DCR.0b013e31829196d0. PMID 23739196